CLINICAL TRIAL: NCT02623582
Title: Pilot Study of RNA-Redirected Autologous T Cells Engineered to Contain Anti-CD123 Linked to TCR and 4-1BB Signaling Domains in Patients With Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: CD123 Redirected Autologous T Cells for AML
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: This study was terminated due to lack of funding.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 823175 - UPCC 04415
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): The first 3 subjects to receive RNA CART123 cells will receive up to 3 doses of RNA CART123 cells, with no lymphodepleting chemotherapy prior to infusion.
  Interventions: Biological: Autologous Anti-CD 123 CAR TCR/4-1BB-expressing T-lymphocytes
- Cohort 2 (Experimental): The remaining 12 subjects of the study will receive up to six IV doses of RNA CART123 cells.
  Subjects in Cohort 2 may be given lymphodepleting chemotherapy 4 days (+/- 1 day) prior to the first CART123 cell infusion (if ALC> 500/uL).
  Lymphodepleting chemotherapy may be repeated before the fourth dose of RNA CART123 cells (if ALC> 500/uL).
  Lymphodepleting chemotherapy includes a single dose of cyclophosphamide (1g/m2) Weight used for dosing will be the weight obtained prior to the apheresis procedure Cell numbers are based on CAR+ cells with CAR expression determined by flow cytometry Based on the product release criteria, at least 20% of the total cells will be RNA CART123 cells.
  Dosing will not be changed for changes in subject weight The indicated doses are +/- 20% to account for manufacturing variability.
  Interventions: Biological: Autologous Anti-CD 123 CAR TCR/4-1BB-expressing T-lymphocytes; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Autologous Anti-CD 123 CAR TCR/4-1BB-expressing T-lymphocytes — Given IV
Drug: Cyclophosphamide — Given IV
  Arms: Cohort 2

SUMMARY:
Pilot open-label study to estimate the feasibility, safety and efficacy of intravenously administered, RNA electroporated autologous T cells expressing anti-CD123 chimeric antigen receptors expressing tandem TCR and 4-1BB (TCR /4-1BB) costimulatory domains (referred to as RNA CART123) in Acute Myeloid Leukemia (AML) subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age or older with AML with no available curative treatment options using currently available therapies
* Subjects must have a suitable stem cell donor available who may donate cells if the subject needs to undergo allogeneic HCT. Donor may be matched or mismatched and must be found to be suitable according to the institution's standard criteria.
* Subjects with second or subsequent relapse, any relapse refractory to salvage, or with persistent disease after at least two lines of therapy.

  a. Subjects with relapsed disease after prior allogeneic HCT (myeloablative or non-myeloablative) will be eligible if they meet all other inclusion criteria and i. Have experienced graft rejection (no evidence of donor cells by STR analysis on 2 occasions separated by at least 1 month), OR: ii. Donor cells are present but there is no active GVHD, subject does not require immunosuppression and is more than 6 months from transplant
* Subjects must have evaluable disease defined as >5% blasts on marrow aspirate or biopsy, extramedullary disease (CNS involvement is prohibited), or at least 20% blasts in the peripheral blood within 2 weeks prior to enrollment. Note: subjects with second or subsequent relapse are considered to have evaluable disease even without meeting the above morphologic criteria if they are found to have persistent recurrent disease-associated molecular or cytogenetic abnormalities.
* Creatinine < 1.6 mg/dl
* ALT/AST must be < 5 x upper limit of normal unless related to disease
* Bilirubin < 2.0 mg/dl, unless subject has Gilbert's syndrome (≤3.0 mg/dL);
* ECOG Performance status 0-2.
* Left ventricular ejection fraction > 40% as confirmed by ECHO/MUGA
* Written informed consent is given.
* Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion criteria:

* Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum pregnancy test at enrollment. A urine pregnancy test will be performed within 48 hours before infusion.
* HIV infection.
* Active hepatitis B or hepatitis C infection.
* Concurrent use of systemic steroids or immunosuppressant medications. Recent or current use of inhaled steroids or physiologic replacement with hydrocortisone is not exclusionary.
* Absolute lymphocyte count <500/uL
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* Subjects with signs or symptoms indicative of CNS involvement. A CNS evaluation should be performed as clinically appropriate to rule out CNS involvement.
* Known history of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
* Class III/IV cardiovascular disability according to the New York Heart Association Classification.
* Patients with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system
* Subjects with clinically apparent arrhythmia, or arrhythmias that are not stable on medical management, within 2 weeks of the Screening/Enrollment visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08-26 (Actual); Study Completion 2016-11-18 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Saar Gill, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes